CLINICAL TRIAL: NCT01852877
Title: Seek, Test, Treat: An Integrated Jail-Prison-Community Model for Illinois
Brief Title: Seek, Test, Treat, Retain: An Integrated Jail-Prison-Community Model for Illinois
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lawrence J. Ouellet, Ph.D., Research Professor, University of Illinois at Chicago
Other Study IDs: 2011-0619; 1R01DA030796 (NIH)
Record Dates: First submitted 2013-05-08; First posted 2013-05-14 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: HIV Infections
Keywords: HIV Diagnosis; Case Management; Telemedicine; Patient Compliance; Prisoners
MeSH Terms: conditions — HIV Infections; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum

GROUPS / COHORTS (2):
- Jail: HIV testing, corrections case mgt: For all jail detainees regardless of HIV status, we observed the uptake of opt-out and opt-in HIV testing. For HIV-positive jail detainees leaving jail, we observed 1) health outcomes for corrections case management versus other than corrections case management, 2) the impact of an incentive to visit an HIV service organization after release from jail
  Interventions: Behavioral: Corrections case management
- Prison: telemed, corrections case mgt: We compared outcomes for for HIV-positive prisoners before and after the implementation of telemedicine to deliver HIV medical care. For HIV-positive prisoners released from prison and returning to Chicago, we observed health outcomes for those enrolled in corrections case management those not enrolled in corrections case management.
  Interventions: Behavioral: Corrections case management

INTERVENTIONS:
Behavioral: Corrections case management — Corrections case management is a long-term (18-24 months) program that seeks to improve the linkage of HIV-positive persons recently released from jail or prison to community-based HIV care, retain them in care, and reduce recidivism. Compared to the long-standing Ryan White case management program, corrections case management has greater access to housing and a greater emphasis on employment. Clients completing the program are then linked to the Ryan White case management program.

SUMMARY:
Aim-1: Evaluate opt-out versus opt-in testing for the human immunodeficiency virus (HIV) at the Cook County jail and the Illinois Department of Corrections Northern Intake facilities. Outcomes of interest include a) uptake of each HIV testing strategy, b) comparative effectiveness of identifying HIV-positive cases, new cases and undisclosed cases, and c) predictors of HIV testing.

Aim-2: Evaluate two case management strategies - "correctional case management" and "transitional case management" - designed to improve linkage and adherence to appropriate medical care after release from incarceration. Correctional case management is a longer-term, more intense approach while transitional case management seeks to meet the clients' immediate needs, link them to Ryan White case management, and then support the Ryan White case manager in assisting these clients. Correctional case management will be compared to the standard of care for jail detainees, and to transitional case management for persons leaving prison. Outcomes of interest include, (a) HIV viral load and CD4 cell counts over time, (b) adherence to medication, and (c) visits to medical providers.

Aim-3: Evaluate the impact of an incentive for HIV-positive detainees released from jail to visit an HIV service organization where they can be linked to medical care and case management. Outcomes of interest are essentially the same as Aim-2.

Aim-4: Assess university-based telemedicine as means to improve care of state prison inmates living with HIV. Outcomes of interest include medication regimens, HIV viral load and CD4 cell counts, and associated health conditions.

Aim-5: Assess the uptake of partner notification and social network HIV counseling and testing involving HIV-positive persons released from jail and prison as a means to extend the reach of the 'seek, test, treat and retain' (STTR) model into the community.

ELIGIBILITY:
Inclusion Criteria:

* For assessing opt-out and opt-in HIV testing: all detainees in Cook County Jail and all prisoners in the Northern Intake facilities of the Illinois Department of Corrections (IDOC)
* For assessing telemedicine: all HIV-positive IDOC prisoners who have received treatment for HIV. -- For assessing case management: all IDOC HIV telemedicine patients who have been released from prison and returned to Chicago in the past 60 days, and all known HIV-positive jail detainees likely to be returning the community (Chicago) within 60 days of contact with the jail's HIV clinic
* For assessing a post-release incentive to visit an HIV service organization, and uptake of post-release partner notification and social network HIV testing: all former detainees participating in the case management evaluation

Exclusion Criteria:

* Less than 18 years old
* Unable to speak English or Spanish
* Incapable of providing informed consent
* For jail detainees: being under extradition to a locale outside Cook County or a high likelihood of being sent to prison rather than being released to the community
* For prison inmates: being under extradition to a locale outside Illinois

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Detainees in Cook County Jail, prisoners in the Illinois Department of Corrections
Sampling Method: Non-Probability Sample
Enrollment: 784 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change in HIV viral load | baseline and 6, 12, 18 months post-baseline

SECONDARY OUTCOMES:
Change in CD4 cell count | baseline and 6, 12, 18 months post-baseline
Change in community-level HIV viral load | baseline and 18 months post-baseline

OTHER OUTCOMES:
Change in adherence to HIV medication | baseline and 6, 12, 18 months post-baseline
Change in visits to HIV medical care provider | baseline and 6, 12, 18 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Ouellet, PhD, Principal Investigator — University of Illinois at Chicago; Jeremy D Young, MD, Principal Investigator — University of Illinois at Chicago; Chad Zawitz, MD, Principal Investigator — Cermak Health Services, Cook County
Locations (3):
- United States (3):
  - Illinois Department of Corrections, Chicago, Illinois
  - University of Illinois at Chicago, School of Public Health, COIP, Chicago, Illinois
  - Cermak Health Services, Cook County Jail, Chicago, Illinois